CLINICAL TRIAL: NCT05986994
Title: Role of microRNAs as Diagnostic and Prognostic Biomarkers of Neonatal Perinatal Asphyxia and Hypoxic Ischemic Encephalopathy
Brief Title: Identification of a Pool of miRNA to Improve Early Management of Perinatal Asphyxia and Hypoxic Ischemic Encephalopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Buon Consiglio Fatebenefratelli (Other)
Collaborators: Federico II University (Other)
Responsible Party: Principal Investigator, Giuseppe De Bernardo, Chief Physician, Ospedale Buon Consiglio Fatebenefratelli
Other Study IDs: 495
Record Dates: First submitted 2023-07-08; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Asphyxia Perinatal
Keywords: newborn; microRNA; asphyxia; encephalopathy; hypothermia
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Asphyxia; Brain Diseases; Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: 15 healthy newborns with umbilical cord arterial pH between 7.26 and 7.35
  Interventions: Diagnostic Test: microRNA
- Group B: 15 newborns with metabolic acidosis at birth with umbilical cord arterial pH at birth < 7.12 and who do not practice therapeutic hypothermia due to lack of enrollment criteria
  Interventions: Other: Metabolic acidosis; Diagnostic Test: microRNA
- Group C: 15 newborns with metabolic acidosis at birth with umbilical cord arterial pH at birth < 7.12 and practicing therapeutic hypothermia in accordance with current guidelines
  Interventions: Other: Metabolic acidosis; Diagnostic Test: microRNA; Other: Hypothermia

INTERVENTIONS:
Other: Metabolic acidosis — Metabolic acidosis at birth with umbilical cord arterial pH at birth < 7.12
  Groups: Group B; Group C
Diagnostic Test: microRNA — Evaluation of microRNA levels
Other: Hypothermia — Therapeutic induced hypothermia refers to a lowering of the central body temperature for therapeutic purposes
  Groups: Group C

SUMMARY:
Hypoxic-ischemic encephalopathy is the most common cause of neurological damage in the neonatal period. It has an incidence of about 1.5-2.5% of livebirths in developed countries. It is associated with a high rate of mortality and morbidity. Major neurological outcomes such as cerebral palsy, mental retardation, learning disabilities, epilepsy occur in approximately 25% of survivors. The diagnostic and prognostic tools currently available for enrollment have limitations and additional reliable biomarkers are needed for all phases of clinical management. Sarnat staging has taken on a role in identifying those infants who may benefit from treatment of hypothermia, resulting in the need for neurological evaluation and staging within 6 hours of life. Therapeutic hypothermia is still the best therapeutic treatment.

A new tool in neuroscience research is represented by micro-ribonucleic acid (microRNA) profiling. The presence of microRNAs in blood, urine and saliva and the ability to measure their levels non-invasively has opened new doors in the search for peripheral biomarkers for the diagnosis and prognosis of neurodegenerative diseases and also as possible pharmacological targets.

The aim of the present study is to analyze a specific cluster of miRNAs selected from data obtained by macroarray (NGS Pannel) on the entire microRNAome in healthy newborns with normal cord arterial pH value (7.26-7.35) as control cases and in newborns with fetal metabolic acidosis with a pH threshold value lower than 7.12 of the blood gas analysis from cord arterial blood. This latter group will be further stratified into two groups, neonates who will practice therapeutic hypothermia according to current guidelines and a further group who will not practice therapeutic hypothermia. This study will make a further international contribution in evaluating and identifying the potential of microRNAs as diagnostic and prognostic biomarkers in perinatal asphyxia and hypoxic ischemic encephalopathy. Furthermore, the study aims to identify specific microRNA sequences as new possible markers to be used as an additional parameter for the enrollment of therapeutic hypothermia, especially in cases of mild hypoxic-ischemic encephalopathy.

DETAILED DESCRIPTION:
Hypoxic-ischemic encephalopathy is the most common cause of neurological damage in the neonatal period. It has an incidence of about 1.5-2.5% of livebirths in developed countries. It is associated with a high rate of mortality and morbidity. About 1 million newborns worldwide die of hypoxic-ischemic encephalopathy. In the neonatal period die between 20 and 50% of asphyxiated infants who develop hypoxic-ischemic encephalopathy. Major neurological outcomes such as cerebral palsy, mental retardation, learning disabilities, epilepsy occur in approximately 25% of survivors. Therapeutic hypothermia is still the best therapeutic treatment. The diagnostic and prognostic tools currently available for enrollment have limitations and additional reliable biomarkers are needed for all phases of clinical management. One of the difficulties in interpretation lies in the identification of mild-grade hypoxic-ischemic encephalopathy which appears to be operator dependent, as well as the timing of the diagnosis. Sarnat staging has taken on a role in identifying those infants who may benefit from treatment of hypothermia, resulting in the need for neurological evaluation and staging within 6 hours of life. This is a relatively short time frame in which it is plausible to think that mild hypoxic-ischemic encephalopathy could become moderate at 6 h. In fact, some studies have retrospectively demonstrated the outcome of infants with mild hypoxic-ischemic encephalopathy defined between 1 and 6 hours of birth showing worse neurodevelopmental outcomes than the data reported in the pre-hypothermia literature.

A new tool in neuroscience research is represented micro-ribonucleic acid (microRNA) profiling. Significant numbers of microRNAs have been observed outside cells including various body fluids. MicroRNAs have been detected in plasma, serum, milk, tears, saliva, urine, amniotic fluid, cerebrospinal fluid, and seminal fluid. Despite the instability of most RNA molecules in the extracellular environment, the presence and apparent stability of microRNAs has proven surprising. In particular, they were found to be very stable and resistant to RNases, freezing and pH variations. The presence of microRNAs in blood, urine and saliva and the ability to measure their levels non-invasively has opened new doors in the search for peripheral biomarkers for the diagnosis and prognosis of neurodegenerative diseases and also as possible pharmacological targets. In view of their usefulness, in recent years more and more different microRNAs have been analyzed as possible diagnostic and prognostic markers of perinatal asphyxia but specific sequences with high specificity and sensitivity have not yet been identified as markers of neonatal hypoxia and hypoxic ischemic encephalopathy with the need to perform further confirmatory studies. The aim of the present study is to analyze a specific cluster of miRNAs selected from data obtained by macroarray (NGS Pannel) on the entire microRNAome in healthy newborns with normal cord arterial pH value (7.26-7.35) as control cases and in newborns with fetal metabolic acidosis with a pH threshold value lower than 7.12 of the blood gas analysis from cord arterial blood. This latter group will be further stratified into two groups, neonates who will practice therapeutic hypothermia according to current guidelines and a further group who will not practice therapeutic hypothermia. This study will make a further international contribution in evaluating and identifying the potential of microRNAs as diagnostic and prognostic biomarkers in perinatal asphyxia and hypoxic ischemic encephalopathy. Furthermore, the study aims to identify specific microRNA sequences as new possible markers to be used as an additional parameter for the enrollment of therapeutic hypothermia, especially in cases of mild hypoxic-ischemic encephalopathy. Subsequently, this study will allow to evaluate their potential as new possible pharmacological targets in the pediatric field for hypoxic-ischemic encephalopathy in future preclinical studies as already reported in the literature in various preclinical studies, as therapeutic perspectives in ischemic stroke in adults.

ELIGIBILITY:
Inclusion Criteria:

* newborns with at least 35 weeks of gestational age
* body weight of at least 1800 g

Exclusion Criteria:

* Withdrawal of informed consent

Ages: 35 Weeks to 42 Weeks | Sex: All
Age Groups: Child
Study Population: All patients transferred to the Buon Consiglio Fatebenefratelli hospital will be eligible
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-07-18 (Estimated); Study Completion 2024-07-18 (Estimated)

PRIMARY OUTCOMES:
Evaluation of microRNA levels | 60 minutes of life
  Quantitative characterization of microRNAs (ng/uL) in healthy neonates and neonates with metabolic acidosis at birth with or without therapeutic hypothermia and who developed hypoxic ischemic encephalopathy
Qualitative evaluation of microRNAs | 60 minutes of life
  Characterization of the type of microRNAs in healthy neonates and neonates with metabolic acidosis at birth with or without therapeutic hypothermia and who developed hypoxic ischemic encephalopathy
Evaluation of microRNA levels | 3 hours of life
  Quantitative characterization of microRNAs (ng/uL) in healthy neonates and neonates with metabolic acidosis at birth with or without therapeutic hypothermia and who developed hypoxic ischemic encephalopathy
Qualitative evaluation of microRNAs | 3 hours of life
  Characterization of the type of microRNAs in healthy neonates and neonates with metabolic acidosis at birth with or without therapeutic hypothermia and who developed hypoxic ischemic encephalopathy
Evaluation of microRNA levels | 72 hours of life
  Quantitative characterization of microRNAs (ng/uL) in healthy neonates and neonates with metabolic acidosis at birth with or without therapeutic hypothermia and who developed hypoxic ischemic encephalopathy
Qualitative evaluation of microRNAs | 72 hours of life
  Characterization of the type of microRNAs in healthy neonates and neonates with metabolic acidosis at birth with or without therapeutic hypothermia and who developed hypoxic ischemic encephalopathy

SECONDARY OUTCOMES:
Predictive role of microRNAs | 60 minutes of life
  To assess the role of microRNAs as marker of perinatal asphyxia
Predictive role of microRNAs | 60 minutes of life
  To assess the role of microRNAs as markers of mild hypoxic ischemic encephalopathy
Predictive role of microRNAs | 3 hours of life
  To assess the role of microRNAs as markers of perinatal asphyxia
Predictive role of microRNAs | 3 hours of life
  To assess the role of microRNAs as markers of mild hypoxic ischemic encephalopathy
Predictive role of microRNAs | 72 hours of life
  To assess the role of microRNAs as markers of perinatal asphyxia
Predictive role of microRNAs | 72 hours of life
  To assess the role of microRNAs as markers of mild hypoxic ischemic encephalopathy

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe De Bernardo, Prof, Principal Investigator — Buon Consiglio Fatebenefratelli Hospital
Locations (2):
- Italy (2):
  - Department of Neuroscience, Reproductive and Dentistry Sciences, University of Naples Federico II, Naples
  - Department of Woman and Child, Buon Consiglio Fatebenefratelli Hospital, Napoli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gunn AJ. Cerebral hypothermia for prevention of brain injury following perinatal asphyxia. Curr Opin Pediatr. 2000 Apr;12(2):111-5. doi: 10.1097/00008480-200004000-00004. PMID 10763759
- [Result] Vinciguerra A, Cepparulo P, Anzilotti S, Cuomo O, Valsecchi V, Amoroso S, Annunziato L, Pignataro G. Remote postconditioning ameliorates stroke damage by preventing let-7a and miR-143 up-regulation. Theranostics. 2020 Oct 27;10(26):12174-12188. doi: 10.7150/thno.48135. eCollection 2020. PMID 33204336
- [Result] DE Bernardo G, Riccitelli M, Giordano M, Toni AL, Sordino D, Trevisanuto D, Buonocore G, Perrone S. Does high fidelity neonatal resuscitation simulation increase salivary cortisol levels of health care providers? Minerva Pediatr (Torino). 2023 Dec;75(6):884-889. doi: 10.23736/S2724-5276.21.05873-0. Epub 2021 Jun 21. PMID 34152109
- [Result] Locci E, Bazzano G, Demontis R, Chighine A, Fanos V, d'Aloja E. Exploring Perinatal Asphyxia by Metabolomics. Metabolites. 2020 Apr 4;10(4):141. doi: 10.3390/metabo10040141. PMID 32260446
- [Result] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Result] De Bernardo G, De Santis R, Giordano M, Sordino D, Buonocore G, Perrone S. Predict respiratory distress syndrome by umbilical cord blood gas analysis in newborns with reassuring Apgar score. Ital J Pediatr. 2020 Feb 12;46(1):20. doi: 10.1186/s13052-020-0786-8. PMID 32050997
- [Result] Hull J, Dodd KL. Falling incidence of hypoxic-ischaemic encephalopathy in term infants. Br J Obstet Gynaecol. 1992 May;99(5):386-91. doi: 10.1111/j.1471-0528.1992.tb13754.x. PMID 1622910
- [Result] Conway JM, Walsh BH, Boylan GB, Murray DM. Mild hypoxic ischaemic encephalopathy and long term neurodevelopmental outcome - A systematic review. Early Hum Dev. 2018 May;120:80-87. doi: 10.1016/j.earlhumdev.2018.02.007. Epub 2018 Feb 26. PMID 29496329
- [Result] O'Sullivan MP, Looney AM, Moloney GM, Finder M, Hallberg B, Clarke G, Boylan GB, Murray DM. Validation of Altered Umbilical Cord Blood MicroRNA Expression in Neonatal Hypoxic-Ischemic Encephalopathy. JAMA Neurol. 2019 Mar 1;76(3):333-341. doi: 10.1001/jamaneurol.2018.4182. PMID 30592487
- [Result] Ponnusamy V, Yip PK. The role of microRNAs in newborn brain development and hypoxic ischaemic encephalopathy. Neuropharmacology. 2019 May 1;149:55-65. doi: 10.1016/j.neuropharm.2018.11.041. Epub 2019 Feb 1. PMID 30716413
- [Result] Walsh BH, Inder TE. MRI as a biomarker for mild neonatal encephalopathy. Early Hum Dev. 2018 May;120:75-79. doi: 10.1016/j.earlhumdev.2018.02.006. Epub 2018 Feb 17. PMID 29463417
- [Result] Weber JA, Baxter DH, Zhang S, Huang DY, Huang KH, Lee MJ, Galas DJ, Wang K. The microRNA spectrum in 12 body fluids. Clin Chem. 2010 Nov;56(11):1733-41. doi: 10.1373/clinchem.2010.147405. Epub 2010 Sep 16. PMID 20847327